CLINICAL TRIAL: NCT02328963
Title: A Multicenter, Two Arms, Randomized, Open Label Clinical Phase IV Study Investigating the Proportion of CMV Seropositive Kidney Transplant Recipients Who Will Develop a CMV Infection Within the First 6 Months Post-transplantation When Treated With an Immunosuppressive Regimen Including Everolimus (Certican®) and Reduced Dose of Cyclosporine A (Neoral®) Versus an Immunosuppressive Regimen With Mycophenolic Acid (Myfortic®) and Standard Dose of Cyclosporine A (Neoral®).
Brief Title: Proportion of CMV Seropositive Kidney Transplant Recipients Who Will Develop a CMV Infection When Treated With an Immunosuppressive Regimen Including Everolimus and Reduced Dose of Cyclosporine Versus an Immunosuppressive Regimen With Mycophenolic Acid and Standard Dose of Cyclosporine A
Acronym: EVERCMV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2012/29
Record Dates: First submitted 2014-09-01; First posted 2014-12-31 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Transplantation Infection; Cytomegalovirus Infection
Keywords: Cytomegalovirus infection and disease; CMV-seropositive recipients; Everolimus; preemptive strategy; mTOR inhibitor
MeSH Terms: conditions — Cytomegalovirus Infections; Disease | interventions — Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Everolimus + reduced dose of cyclosporine A
  Interventions: Drug: Everolimus
- mycophenolic acid (Active Comparator): mycophenolic acid + standard dose of cyclosporin A
  Interventions: Drug: mycophenolic acid

INTERVENTIONS:
Drug: Everolimus — Everolimus : 0.75 bid, targeted to 3-8 ng/ml
  Cyclosporin A :
  CsA target ranges for Arm 1 will be 100-200 ng/mL from Day 3 to Month 2, decreasing to 75-150 ng/mL from Month 2 to Month 4 and 25-50 ng/mL from Months 6 to 12.
  Corticosteroids :
  Méthylprednisolone: 500 mg at Day 0, 120 mg à Day 1. Prednisone or equivalent: 20 mg/d from Day 3. Corticosteroid dosing will be tapered according to center standard practice but to not less than 5 mg per day for the duration of the 12-month study
  Basiliximab :Day 0: 20 mg ; Day 4: 20 mg
  Arms: Everolimus
Drug: mycophenolic acid — Mycophenolic acid :
  1080 mg bid for one month, then 720 mg bid
  Cyclosporin A :
  CsA target ranges for Arm 1 will be 100-200 ng/mL from Day 3 to Month 2, decreasing to 75-150 ng/mL from Month 2 to Month 4 and 25-50 ng/mL from Months 6 to 12.
  Corticosteroids :
  Méthylprednisolone: 500 mg at Day 0, 120 mg à Day 1. Prednisone or equivalent: 20 mg/d from Day 3. Corticosteroid dosing will be tapered according to center standard practice but to not less than 5 mg per day for the duration of the 12-month study
  Basiliximab :Day 0: 20 mg ; Day 4: 20 mg
  Arms: mycophenolic acid

SUMMARY:
Cytomegalovirus (CMV) infection is the most frequent opportunistic viral infection after transplantation. It is associated with an increased incidence of acute rejection and lower graft and patient survivals. The goal of this study is to demonstrate that an immunosuppressive regimen associating everolimus and reduced dose of cyclosporine A can prevent acute rejection episodes as efficiently as standard regimen but also efficiently reduce the incidence of CMV infection at 6 months post-transplantation.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection is the most frequent opportunistic viral infection after kidney transplantation. Therefore most of the patients receive an universal prophylaxis. On the contrary to CMV naïve patients, seropositive recipients (R+) have already mounted a specific immunologic response directed against the virus, which is not completely abrogated by immunosuppressive drugs. Although CMV infection management guidelines offer little guidance on immunosuppressive therapy for preventing CMV infection and disease, recent data plead for reappraising the place of mTOR inhibitors in this situation. The potential anti-CMV action of these molecules could be added to their potential antitumor effect and their equivalent immunosuppressive efficacy in kidney transplant recipients at low immunological risk. By the way, it could represent an alternative of a systematic universal prophylaxis in R+ kidney transplant recipients. However, the proof of this anti-CMV action must be confirmed in vivo in a study, which could have a close monitoring of CMV infection.

We therefore designed a prospective multicentric randomized controlled trial comparing an immunosuppressive regimen based on everolimus and reduced dose of cyclosporine A to a regimen based on mycophenolic acid and standard dose of cyclosporine A, in order to demonstrate the superiority of the first one in the prevention of CMV infection.

Subjects will be randomized to one of the two treatment arms and will be followed for a period of 12 months. Whole blood CMV real time PCR will be performed every week during the first three months, then every two weeks from Month 3 to Month 6, then at Months 8, 10 and 12. Incidence of CMV infection will be compared between the two arms at 6 and 12 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* End stage kidney disease and a suitable candidate for primary renal transplantation or re-transplantation.
* Patient seropositive for CMV (confirmed within two weeks post-transplant) and having received an allograft from a CMV seropositive or seronegative donor.
* Receiving a kidney transplant from a deceased or living donor with compatible ABO blood type.
* Female subject of childbearing potential must have a negative serum pregnancy test at enrollment and must agree to maintain effective birth control during the study and two months later the discontinuation of the test drug.
* Total ischemia time below 36 hours.
* Capable of understanding the purpose and risks of the study.
* Fully informed and having given written informed consent (signed Informed Consent has been obtained).
* Affiliation to the social security regimen

Exclusion Criteria:

* CMV seronegative patient.
* Historical or current TGI (French equivalence of calculated PRA) > 85 %
* Presence of historical or current anti-HLA donor specific antibodies
* Patient who received anti-CMV therapy within the past 30 days prior to screening.
* Receiving or having previously received an organ transplant other than a kidney.
* Receiving a graft from a non-heart-beating donor.
* Patient known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B (HBV; HBs Ag positive) or Hepatitis C (HCV; anti-HCV Ab positive).elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin levels ≥ 2 times the upper value of the normal range of the investigational site or receiving a graft from a hepatitis C or B positive donor.
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer.
* Known allergy or intolerance to everolimus, valganciclovir, ganciclovir, mycophenolic acid, basiliximab, corticosteroids, or cyclosporine A or any of the product excipients.
* Severe hyperlipidemia defined by: total cholestérol ≥ 9,1 mmol/L (≥ 350 mg/dL) et/ou triglycérides ≥ 8,5 mmol/l (≥ 750 mg/dL) in spite an adequate medication.
* Patient has adequate hematological post-transplant defined as:

  1. Absolute neutrophil count (ANC) > 1000 cells/μL.
  2. Platelet count > 50,000 cells/μL.
  3. Hemoglobin > 8.0 g/dL.
* Requiring initial therapy with induction immunosuppressive antibody preparations, such as anti-thymocyte globulins or rituximab or IVIG.
* Currently participating in another clinical trial investigating drugs. Observational studies are not considered as an exclusion criteria
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator.
* Unlikely to comply with the visits scheduled in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Number of participants without CMV infection and without graft loss in CMV seropositive kidney transplant recipients. | 6 months post-transplantation
  The primary objective of this study is to compare the survival without CMV infection and without graft loss in CMV seropositive kidney transplant recipients, within the first 6 months post-transplantation when treated with an immunosuppressive regimen including everolimus (Certican®) and reduced dose (RD) of cyclosporine A (Néoral®) versus an immunosuppressive regimen with mycophenolic acid (Myfortic®) and standard dose (SD) of cyclosporine A (Néoral®).

SECONDARY OUTCOMES:
Proportion of patients who will develop CMV disease | 6 and 12 months post-transplantation
  The proportion of patients who will develop CMV disease during the first 6 and 12 months post-transplantation (CMV disease includes both CMV syndrome and CMV tissue-invasive disease).
Proportion of patient with graft loss, death and loss of follow-up | 12 months post-transplantation
Proportion of patient with acute rejection, graft loss, death and loss of follow-u | 12 months
Level to the first CMV DNAemia | Throughout the study
Time to the first CMV disease | Throughout the study
Proportion of patients treated for CMV infection in both groups | 6 months
Half-life of decreasing of DNAemia | after initiation of anti-CMV therapy
Occurrence of treatment failure, defined as the absence of viral eradication. | Day 49 (or 8 weeks) after the initiation of anti-CMV therapy
Occurrence of CMV mutation (UL97 ou UL54) associated with a resistance to an anti-CMV therapy. | Throughout the study
Graft function | 6 and 12 months post-transplantation
  Graft function defined as glomerular filtration rate (GFR) estimated by simplified MDRD formula and proteinuria/creatininuria ratio.
Proportion of patients with biopsy-proven acute rejection (BPAR) | 6 and 12 months post-transplantation
Degree of interstitial fibrosis/tubular atrophy | 12 months on protocol biopsies
Graft and patient survival | 6 and 12 months post-transplantation
Proportion of BK virus viremia | month 1, 3, 6 and 12
Proportion of patients with adverse events (AE) and/or serious adverse events (SAE) including opportunistic infections and neoplasias. | 12 months
Proportion of patients with haematological disorders | 12 months
  The proportion of patients with haematological disorders (neutropenia, anaemia, thrombopenia)
Proportion of patients with diarrhea | 12 months
Proportion of dyslipidemia | 12 months
Proportion of patients with occurrence of New Onset Diabetes Mellitus as defined by American Diabetic Association (ADA) criteria. | 12 months
Proportion of patients who will discontinue the immunosuppressive treatment and the reasons why. | 12 months
Proportion of patients with delayed graft function | 12 months
Proportion of lymphocele | 12 months
Time to the first CMV DNAemia | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Lionel COUZI, MD, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - CHU La Cavale Blanche, Brest
  - CHRU Caen - Hôpital de Caen, Caen
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - APHP - Hôpital Necker, Paris
  - APHP - Kremlin Bicetre, Paris
  - CHRU Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse

REFERENCES:
- [Derived] Kaminski H, Marseres G, Yared N, Nokin MJ, Pitard V, Zouine A, Garrigue I, Loizon S, Capone M, Gauthereau X, Mamani-Matsuda M, Coueron R, Duran RV, Pinson B, Pellegrin I, Thiebaut R, Couzi L, Merville P, Dechanet-Merville J. mTOR Inhibitors Prevent CMV Infection through the Restoration of Functional alphabeta and gammadelta T cells in Kidney Transplantation. J Am Soc Nephrol. 2022 Jan;33(1):121-137. doi: 10.1681/ASN.2020121753. Epub 2021 Nov 1. PMID 34725108